CLINICAL TRIAL: NCT03454620
Title: Phase 1b/2a Study of GC1118 in Combination With Irinotecan or FOLFIRI in Patients With Recurrent/Metastatic Solid Tumor
Brief Title: A Study to Assess Safety, Efficacy, Immunogenicity, PK of GC1118 With Combination Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC1118_P12
Record Dates: First submitted 2018-02-13; First posted 2018-03-06 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer; Solid Tumor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC1118 combination with irinotecan (Experimental): GC1118 weekly(3mg or 4mg) + irinotecan 180mg/m2 biweekly dosing
  Interventions: Drug: irinotecan
- GC1118 combination with FOLFIRI (Experimental): GC1118 weekly(3mg or 4mg) + FOLFIRI biweekly dosing
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: irinotecan — GC1118 combination with irinotecan
  Arms: GC1118 combination with irinotecan
Drug: FOLFIRI — GC1118 combination with FOLFIRI
  Arms: GC1118 combination with FOLFIRI

SUMMARY:
The purpose of the study is to assess the safety and tolerability of GC1118 in combination with irinotecan or FOLFIRI in order to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D)

DETAILED DESCRIPTION:
A Phse 1b/2a, dose-finding, open-label, prospective study

This study consists of the Phase 1b part designed to determine the MTD and RP2D of GC1118 when administered in combination with irinotecan or FOLFIRI to patients with recurrent metastatic solid tumors and the Phase 2a part designed to assess the efficacy of GC1118 in combination with FOLFIRI as second-line therapy for recurrent/metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1b: Histologically or cytologically confirmed recurrent/metastatic solid cancer patients with no available standard treatment and be expected to have the anti-tumor effect with combination of GC1118 and irinotecan or GC1118 and FOLFIRI by investigator's judgement Phase 2a: Historically or cytologically confirmed, 1) EGFR-positive, KRAS/NRAS and BRAF wild type recurrent/metastatic colorectal cancer patients who failed first line chemo or targeted therapies (fluoropyrimidine-based or oxaliplatin containing chemotherapy) or whose disease were progressed within 6 months after the last dose of above mentioned treatments; Disease progression during treatment or within 6 months after completion of adjuvant/neoadjuvant chemotherapy is also considered as first line treatment failure 2) Medically documented non-HER2 overexpression (HER2 3+ or HER2+/FISH+) and EGFR 2+ or 3+ expressing recurrent/metastatic gastric cancer patients who failed (radiologically progressed) second line chemo or targeted therapies
2. Male of female, 19 years of age or older
3. ECOS PS 0 or 1
4. Life expectancy of 3 months or longer
5. Phase 2a: Presence of at least one measurable lesion according to the RECIST criteria v1.1
6. Phase 2a: Demonstration of each cohort requirements including EGFR positive, KRAS/NRAS and BRAF wild type, EGFR 2+ or 3+ expression, and etc.
7. Adequate bone marrow function, renal function, and hepatic function
8. All AEs caused by previous anticancer therapies, including surgery, chemotherapy, and radiation therapy,have recovered to CTCAE grade 1 or below (except alopecia)

Exclusion Criteria:

1. Any of the following medical histories 1) Major surgery, open biopsy, or significant traumatic injury within 4 weeks prior to the first investigational products administration or adverse events are not resolved from such procedure or injury 2) Other malignancies (exception; any of the following status are eligible) i. Disease free for 3 years or completely resected non-melanoma skin cancer ii. Successfully treated in carcinoma in situ (CIS) iii. Ta, CIS, or T1a staged superficial bladder cancer which is completely cured iv. Papillary thyroid cancer which is not being progressed without ongoing treatment v. Prostate cancer which is surgically or medically cured and is not likely to recur within 2 years
2. Any of the following concurrent disease 1) Known brain metastasis 2) Active infection requiring systemic anti-microbial therapy 3) Human immunodeficiency virus infection or active hepatitis B or C 4) Chronic inflammatory bowel disease 5) Clinically significant interstitial lung disease or pulmonary fibrosis 6) Clinically significant hepatic disease including decompensated liver cirrhosis, etc
3. Any of the following medication histories 1) Phase 2a recurrent/metastatic colorectal cancer: Treated with irinotecan containing regimen as first line treatment for recurrent/metastatic cancer 2) Phase 2a: Prior EGFR targeting antibody therapy 3) Received chemotherapy, immunotherapy, hormone therapy, radiotherapy within 3 weeks (within 6 weeks in case of nitrosourea or mitomycin-c) prior to first investigational products administration (In phase 2, radiotherapy within 3 weeks is not restricted unless the site is measurable lesion) 4) Ongoing or requiring the prohibited medications including immunotherapy, chemotherapy, hormone therapy, or etc. 5) Received other investigational drugs with 4 weeks prior to this investigational products adminstration
4. Medically or psychologically inappropriate conditions for study participation by investigator's judgment
5. Contraindication for FOLFIRI (or irinotecan) therapy
6. Pregnant, possibly pregnant, or lactating women (Women of child bearing potential must test negative for pregnancy within 3 days prior to Cycle1 Day1
7. Refusal to use the following appropriate contraceptives during the clinical study period and for 6 months after the last adminstration of investigational products 1) Implanted intrauterine device or intrauterine system 2) Double barrier methods (Both of condom (for mate) and diaphragm, vaginal sponge, or cervical cap (for female) should be used with spermicide) 3) Surgical sterilization (vasectomy, tubal ligation, etc.)
8. Any other inappropriate conditions for study participation at investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | through study completion, approximately 5 months
  Profile of DLT

SECONDARY OUTCOMES:
Tumor response according to RECIST 1.1 criteria | before start of treatment, every 6 weeks for the duration of treatment, up to approximately 2 years.
  best overall response (BOR)
Tumor response according to RECIST 1.1 criteria | before start of treatment, every 6 weeks for the duration of treatment, up to approximately 2 years.
  objective response rate (ORR)
Pharmacokinetics of GC1118 | through study completion, approximately 5 months
  area under th curve (AUC)
Pharmacokinetics of GC1118 | through study completion, approximately 5 months
  half life
Pharmacokinetics of GC1118 | through study completion, approximately 5 months
  clearance
Pharmacokinetics of GC1118 | through study completion, approximately 5 months
  peak serum concentration (Cmax)
Immunogenicity of GC1118 | every odd number cycles through treatment period, 28 days after the last treatment
  occurrence frequency of anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Yung Jue Bang, M.D.,Ph.D., Principal Investigator — Seoul National University Hosipital
Locations (6):
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeonam
  - Seoul Asan Medical Center, Seoul
  - Seoul National Universtiy Hosipital, Seoul
  - Yonsei University Health Care System, Seoul

IPD SHARING:
Plan to Share IPD: No